CLINICAL TRIAL: NCT00293202
Title: The Effect of Etanercept in Suppression of the Systemic Inflammatory Response in Hemodialysis Patients
Brief Title: Safety and Efficacy Study of the Effect of Etanercept in Hemodialysis Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: We were unable to recruit sufficient patients within the confines of our budget considering the restrains on our recruitment criteria
Sponsor: Kaysen, George A., M.D., Ph.D. (Other)
Collaborators: Amgen (Industry); Dialysis Clinic, Inc. (Industry)
Responsible Party: Principal Investigator, George A. Kaysen, M.D., Ph.D., Professor, Kaysen, George A., M.D., Ph.D.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 200311904
Record Dates: First submitted 2006-02-15; First posted 2006-02-17 (Estimated); Results first posted 2021-05-28 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: End Stage Renal Disease
Keywords: etanercept; malnutrition; inflammation; hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Malnutrition; Inflammation | interventions — Etanercept; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This is a double blind study- one group received 25mg Etanercept twice per week; the other is control - receiving saline twice per week
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Blind Study

ARMS (2):
- Etanercept 25 mg (Active Comparator): Etanercept 25 mg injection twice a week
  Interventions: Drug: Etanercept
- Saline (Placebo Comparator): Saline injection twice a week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etanercept — Hemodialysis patients will receive Etanercept at a dose of 25 mg by subcutaneous injection twice a week
  Other Names: Enbrel
  Arms: Etanercept 25 mg
Drug: Placebo — Hemodialysis patients will receive Saline by subcutaneous injection twice a week
  Other Names: Saline
  Arms: Saline

SUMMARY:
Etanercept is a novel anti-inflammatory agent currently used in patients with rheumatoid arthritis. We are examining whether Etanercept is effective in improving the nutritional status of hemodialysis patients as a consequence of its ability to decrease inflammation.

DETAILED DESCRIPTION:
Hemodialysis patients with end stage renal disease have a high mortality rate. In individual patients, mortality is associated with a low serum albumin concentration, a marker of poor nutritional status, and with elevated C-reactive protein, a marker of inflammation. Since efforts to improve nutrition through dietary intake have not been successful, inflammation is thought to play a key role in determining nutritional status. Recently, it has been shown that malnutrition, inflammation, and atherosclerosis are closely related in patients with chronic renal failure. It is our hypothesis that suppression of the cycle of inflammation, malnutrition, and vascular injury caused by atherosclerosis will improve survival in dialysis patients. This study is designed to examine whether suppression of the inflammatory response can be accomplished safely with Etanercept and to determine if this suppression will improve nutritional status and clinical outcome in hemodialysis patients with poor nutritional status and evidence of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Presence of end stage renal disease

Exclusion Criteria:

* History of Tuberculosis History of Recurrent Infection Recent AMI, Cancer within previous 5 years Presence of Hepatitis B, Hepatitis C, HIV, systemic lupus erythematosis, presence of transcutaneous access (external catheter)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2008-03 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Kaysen, MD, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Medical Center, Sacramento, California, United States

REFERENCES:
- [Result] Don BR, Kim K, Li J, Dwyer T, Alexander F, Kaysen GA. The effect of etanercept on suppression of the systemic inflammatory response in chronic hemodialysis patients. Clin Nephrol. 2010 Jun;73(6):431-8. doi: 10.5414/cnp73431. PMID 20497755
- See also: B.R. Don, K.Kim, J. Li, T. Dwyer, F. Alexander and G.A. Kaysen.The effect of etanercept on suppression of the systemic inflammatory response in chronic hemodialysis patients. 2010; 73: 431-438. doi: 10.5414/CNP73431 — https://pubmed.ncbi.nlm.nih.gov/20497755/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The protocol was approved by the Human Subjects Review Committee of the University of California Davis Medical Center and Dialysis Clinics, Incorporated. Screening started in January 2005, and had to be terminated early due to low enrollment in December 2006
Pre-assignment Details: Subject was consented and screened for safety. Then they have to qualify for 3 monthly screening values. Once deemed qualified for the study, subject then randomized into a double-blind study; to follow regimen of protocols and followed to 52 weeks of study.
Groups:
- Etanercept: Active Comparator: Etanercept 25 mg injection twice a week
  1. 5 Hemodialysis patients will receive Etanercept at a dose of 25 mg by subcutaneous injection twice a week
  2. Do not have active infections
  3. Patient will be followed for 52 weeks
- Placebo: Placebo comparator: Saline injection twice a week
  1. 5 Hemodialysis patients will receive Saline by subcutaneous injection twice a week
  2. Do not have active infections
  3. Patient will be followed for 52 weeks
Period: Overall Study
Arm/Group | Etanercept | Placebo
Started | 5 | 5
Completed | 2 | 3
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — positive ANA (antinuclear antibody) | 1 | 0
Not completed — on-hold due to fistula maturation time | 1 | 0

BASELINE CHARACTERISTICS:
Population: Total number of participant in each group
Groups:
- Etanercept: Etanercept 25 mg injection twice a week
  Etanercept: Hemodialysis patients will receive Etanercept at a dose of 25 mg by subcutaneous injection twice a week
- Placebo: Saline injection twice a week
  Placebo: Hemodialysis patients will receive Saline by subcutaneous injection twice a week
- Total: Total of all reporting groups
Arm/Group | Etanercept | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 1 | 2 | 3
Age, Continuous [Median (Standard Deviation); unit: years] | 51 (16.739) | 55 (15.209) | 53 (15.101)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: Participant]
  United States | 5 | 5 | 10
C-Reactive Protein (CRP) [Mean (Standard Deviation); unit: mg/L] — C-Reactive Protein is serum protein measured in milligram per liter (mg/L). Increase number indicate higher level of inflammation
  mg/L | 29.05 (15.60) | 10.98 (3.95) | 15.79 (28.13)
Albumin [Mean (Standard Deviation); unit: g/dL] — Serum Albumin is measured in gram per deciliter (g/dL). Increase number is a measured of better nutritional status
  g/dL | 3.39 (0.24) | 3.31 (0.21) | 3.37 (0.20)

OUTCOME MEASURES:

1. Primary Outcome: Albumin
Description: An increased serum albumin (ALB) concentration expected. Higher concentrations of Albumin indicate better outcome. Normal ranges of Albumin in this study is from 3.5 to 5.5 gram per deciliter (g/dL). We expect ALB to remain or increase in this study.
Time Frame: 52 weeks
Population: Hemodialysis patients have a high mortality rate caused by poor nutrition and inflammation. The hypothesis is that suppression of inflammation reverses the malnutrition-inflammation syndrome in hemodialysis patients. Etanercept is an anti-inflammatory agent. Thus it is expected that participant given Etanercept will have a reduced amount of inflammation in their bodies and have better nutritional status - indicated by an increase/steady Albumin level.
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- Etanercept: Active comparator: Etanercept 25 mg injection twice a week
  Hemodialysis patients will receive Etanercept at a dose of 25 mg by subcutaneous injection twice a week for a total of 52 weeks.
- Placebo: No Drug: Saline injection twice a week
  Hemodialysis patients will receive Saline by subcutaneous injection twice a week for a total of 52 weeks
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 5 | 5
g/dL | 3.34 (0.22) | 3.42 (0.25)

2. Primary Outcome: C-reactive Protein
Description: A reduced C-reactive protein (CRP) concentration is expected.
Time Frame: 52 weeks
Population: Malnutrition, inflammation, and atherosclerosis affect patients with chronic renal failure. High C-reactive protein is a marker of inflammation. This study is designed to examine whether suppression of the inflammatory response can be accomplished safely with Etanercept. For those who has high CRP level, we expect that CRP level will be reduced
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Placebo: No Drug - Saline injection twice a week
  Hemodialysis patients will receive Saline by subcutaneous injection twice a week for a total of 52 weeks
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 5 | 5
mg/L | 28.96 (26.00) | 11.94 (13.53)

3. Secondary Outcome: Prealbumin (mg/dL)
Description: Effect of treatment on prealbumin (PAB) concentration
Time Frame: 52 weeks
Population: Serum Prealbumin is measured in milligram per deciliter (mg/dL). Increase number is a measured of better nutritional status.
  In the etanercept group we would expect fewer decreases in prealbumin. Decreased level of prealbumin may indicate inflammations may be occurring in the body.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Etanercept 25 mg | Saline
Number analyzed (Participants) | 5 | 5
mg/dL | 32.36 (8.64) | 31.43 (8.83)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse Event collected was in the same category as defined
Arm/Group | Etanercept | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 3/5
Other Adverse Events (participants affected / at risk) | 1/5 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept (N=5) | Placebo (N=5)
Epigastric pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Nausea, vomiting, constipation, and epigastric pain initially thought to be pancreatitis, but later found to be either gastroenteritis or peptic ulcer disease -Not related to Study
Stroke (Nervous system disorders) | 0 (0) | 1 (1) — Stroke, considered related to elective catheterization to evaluate for kidney transplant, due to development of memory loss and left leg weakness (following ventricular fibrillation during catheterization) -not related to Study
CABG (Cardiac disorders) | 0 (0) | 1 (1) — Coronary artery disease syndrome resulting in 3-vessel CABG - not related to Study
Ventricular Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) — Ventricular fibrillation during elective cardiac catheterization for kidney transplant evaluation - Not related to Study
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept (N=5) | Placebo (N=5)
Skin pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Burning pain in hands -Not related to Study
Cold symptoms (General disorders) | 0 (0) | 1 (1) — Fever, cough, chest congestion -Unlikely related to Study
Hematuria, chest pain, nausea and vomiting (General disorders) | 1 (1) | 0 (0) — Hematuria, chest pain, nausea and vomiting - Not related to Study

LIMITATIONS AND CAVEATS:
Only 10 out of 40 subjects recruited. Only 5 out of 10 subject randomized completed the study. The study has been slow to accrue patients due to the large number and stringent inclusion and exclusion criteria so as to optimize safety. This is due to Etanercept as an anti-inflammatory agent that acts directly on a key regulatory protein in the immune system, tumor necrosis factor α. Extreme stringency was intended to prevent the potential unmasking of latent infection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/02/NCT00293202/SAP_000.pdf